CLINICAL TRIAL: NCT06563817
Title: A Prospective, Multi-center, Open-label Study to Observe the Efficacy and Safety of Rapamycin in the Treatment of Communicating Hydrocephalus Secondary to Intraventricular Hemorrhage
Brief Title: The Safety and Efficacy of Rapamycin on Communicating Hydrocephalus Secondary to Intraventricular Hemorrhage
Acronym: Saturn
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-A-2024025
Record Dates: First submitted 2024-08-09; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Communicating Hydrocephalus; Cerebral Intraventricular Hemorrhage; Secondary Normal Pressure Hydrocephalus; Post Hemorrhagic Hydrocephalus
Keywords: Communicating Hydrocephalus; Cerebral Intraventricular Hemorrhage; Rapamycin; Secondary Normal Pressure Hydrocephalus; Post Hemorrhagic Hydrocephalus
MeSH Terms: conditions — Hydrocephalus; Cerebral Intraventricular Hemorrhage | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: All enrolled patients receive treatment with sirolimus (rapamycin), administered in capsule form at a dosage of 0.5 mg per capsule. The capsules, provided by North China Pharmaceutical under the trade name Yixinke, were stored at room temperature. The prescribed regimen involved a daily oral dosage of 1.5 mg for a duration of four weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapamycin treatment group (Experimental): All enrolled patients receive treatment with sirolimus (rapamycin), administered in capsule form at a dosage of 0.5 mg per capsule. The capsules, provided by North China Pharmaceutical under the trade name Yixinke, were stored at room temperature. The prescribed regimen involved a daily oral dosage of 1.5 mg for a duration of four weeks.
  Sirolimus (rapamycin) bioavailability can be affected by food, based on preliminary results of prior drug use. To maintain consistent blood drug concentrations, sirolimus should be taken with or without food on a constant basis. Grapefruit juice slows CYP3A4-mediated metabolism of sirolimus and potentially enhances P-gp-mediated retrograde transport of sirolimus from the small intestinal epithelium to the intestinal lumen. Therefore, it should not be consumed concurrently with sirolimus.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — All enrolled patients receive treatment with sirolimus (rapamycin)#The prescribed regimen involved a daily oral dosage of 1.5 mg for a duration of four weeks.
  Other Names: Sirolimus

SUMMARY:
This prospective, multicenter, open-label clinical trial is designed to evaluate the safety and efficacy of rapamycin in the treatment of communicating hydrocephalus secondary to intraventricular hemorrhage. Additionally, the underlying pathogenic mechanisms associated with this particular type of hydrocephalus will be investigated in greater depth, and populations that may benefit from rapamycin therapy will be identified.

DETAILED DESCRIPTION:
Communicating hydrocephalus secondary to intraventricular hemorrhage is a serious neurological disorder with the main clinical manifestations of ventricular dilatation, gait disturbance, cognitive dysfunction, and urinary incontinence. At present, the sole treatment option for these patients is cerebrospinal fluid shunting. However, complications resulting from this therapy have necessitated multiple surgeries for some patients, which has a significant impact on their quality of life and financial resources. However, recent studies have identified the PI3K-AKT-mTOR pathway as a key contributor to the sequelae of hemorrhagic hydrocephalus. Furthermore, these studies demonstrated that rapamycin, an inhibitor of the PI3K-AKT-mTOR pathway, inhibited cerebrospinal fluid secretion and ventricular dilation in an animal model of hemorrhagic hydrocephalus sequelae. In light of these findings, we propose a prospective, multicenter, open-label clinical trial to evaluate the efficacy and safety of rapamycin in the treatment of communicating hydrocephalus secondary to intraventricular hemorrhage.

The study design was that of a prospective, multicenter, open-label clinical trial. All patients were administered sirolimus (rapamycin) in a dosage of 0.5 mg per capsule. The capsules were provided by the North China Pharmaceutical Company and were stored at room temperature. The treatment course was four weeks, with a dosage of 1.5 mg orally per day. Efficacy and adverse effects were assessed at two weeks, four weeks, the end of treatment, and 12 weeks after the end of treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ventricular dilatation due to intraventricular hemorrhage who clinically present with any one or more of new gait disturbances, cognitive deficits, and urinary incontinence after remission of intraventricular hemorrhage symptoms, and whose brain imaging shows an Evans index (EI) of ≥0.3
2. Age ≥ 18 years and ≤ 70 years
3. Signed informed consent form

Exclusion Criteria:

1. Participation in another medical trial
2. Have other disease that may affect the patient's symptoms (including gait disturbance, cognitive impairment, urinary incontinence)
3. Allergy to the investigational drug
4. Reduced liver function (increased INR or alanine transaminase concentrations in plasma elevated more than 1.5 times reference values)
5. Reduced kidney function with GFR < 50
6. Concomitant treatment with strong CYP3A4/5 inducers or inhibitors, such as diltiazem, ketoconazole, or rifampicin.
7. Active or uncontrolled chronic infection
8. Women who are pregnant or breastfeeding
9. Patients who are bedridden or require urinary catheters for extended periods of time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The objective remission rate of rapamycin for 4 weeks in the treatment of communicating hydrocephalus secondary to intraventricular hemorrhage is evaluated using the Idiopathic Normal Pressure Hydrocephalus Grading Scale (IPNHGS). | From the commencement of treatment to 4 weeks
  Disease relief: Improvement of >1 point on the Idiopathic Normal Pressure Hydrocephalus Grading Scale (iPNHGS) in patients after four weeks of rapamycin treatment compared to pre-treatment.
  Objective remission rate: The ratio of the number of patients who have achieved disease remission to the total number of patients enrolled in the study.

SECONDARY OUTCOMES:
Assessment of the incidence and severity of adverse events, serious adverse events, and other safety parameters (e.g., abnormal laboratory results) based on CTCAE V5.0 | From the commencement of treatment to 12 weeks after discontinuation of dosing
  All events are determined based on CTCAE V5.0
The objective remission rate of rapamycin treatment of communicating hydrocephalus secondary to intraventricular hemorrhage is evaluated using the Idiopathic Normal Pressure Hydrocephalus Grading Scale (IPNHGS). | From the commencement of treatment to 2 weeks of dosing and 12 weeks after discontinuation of dosing
  Disease relief: Improvement of >1 point on the Idiopathic Normal Pressure Hydrocephalus Grading Scale (iPNHGS) in patients after four weeks of rapamycin treatment compared to pre-treatment.
  Objective remission rate: The ratio of the number of patients who have achieved disease remission to the total number of patients enrolled in the study.
The objective remission rates of 3 clinical domains is evaluated using the Idiopathic Normal Pressure Hydrocephalus Grading Scale (IPNHGS). | From the commencement to 2 weeks of dosing, 4 weeks of dosing and 12 weeks after discontinuation of dosing
  The 3 clinical domains include: gait, urinary incontinence, and cognition. For gait, positive outcome was defined that improvement of >1 point in the gait section of iNPHGS; for urinary incontinence, a positive outcome was defined that improvement of >1 point in the urinary section of iNPHGS; For cognition, positive outcome was defined that improvement of >1 point in the cognition section of iNPHGS
Changes in plasma biomarkers | From the commencement to 2 weeks of dosing, 4 weeks of dosing and 12 weeks after discontinuation of dosing
  Change in plasma levels of TNF-α, IL-1β, IL-6, IL-10, IL-8 and IL-2R.
Change in CSF biomarkers | From the commencement to 2 weeks of dosing, 4 weeks of dosing and 12 weeks after discontinuation of dosing
  Change in plasma levels of TNF-α, IL-1β, IL-6, IL-10, IL-8 and IL-2R.
Change in Euro-Quality of Life-5 dimension-5L (EQ-5D-5L) descriptive system | From the commencement to 2 weeks of dosing, 4 weeks of dosing and 12 weeks after discontinuation of dosing
  Measured using EQ-5D-5L using the descriptive system.

OTHER OUTCOMES:
Screening of potential beneficiary population | From the commencement of treatment to 4 weeks
  Identification of a patient population with secondary communicating hydrocephalus after intraventricular hemorrhage that may benefit from rapamycin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Runfa Tian, MD, Study Director — Beijing Tiantan Hospital; Guoyi Gao, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robert SM, Reeves BC, Kiziltug E, Duy PQ, Karimy JK, Mansuri MS, Marlier A, Allington G, Greenberg ABW, DeSpenza T Jr, Singh AK, Zeng X, Mekbib KY, Kundishora AJ, Nelson-Williams C, Hao LT, Zhang J, Lam TT, Wilson R, Butler WE, Diluna ML, Feinberg P, Schafer DP, Movahedi K, Tannenbaum A, Koundal S, Chen X, Benveniste H, Limbrick DD Jr, Schiff SJ, Carter BS, Gunel M, Simard JM, Lifton RP, Alper SL, Delpire E, Kahle KT. The choroid plexus links innate immunity to CSF dysregulation in hydrocephalus. Cell. 2023 Feb 16;186(4):764-785.e21. doi: 10.1016/j.cell.2023.01.017. PMID 36803604